CLINICAL TRIAL: NCT01299207
Title: PITT PCI Xience Registry: A Prospective Evaluation of Dual Antiplatelet Therapy Compliance and Outcomes After Treatment With the Xience Stent
Brief Title: PITT PCI Xience Registry
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Oscar Marroquin, Study Principal Investigator, University of Pittsburgh
Other Study IDs: 0022189
Record Dates: First submitted 2011-02-15; First posted 2011-02-18 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2016-01

CONDITIONS: Coronary Artery Disease
Keywords: Stents; Drug-Eluting Stents; Stent Thrombosis; Bleeding; Dual-Antiplatelet Therapy
MeSH Terms: conditions — Coronary Artery Disease; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CAD treated with Xience stents: Patients with CAD who undergo successful stenting with the Xience drug-eluting stent will represent the patient population.

SUMMARY:
Stents are devices utilized to treat cholesterol blockages of the coronary (heart) arteries. The introduction of drug-eluting (coated) stents into clinical practice is regarded as a revolutionary breaktrhough, as it has reduced the incidence of re-narrowing of the arteries after percutaneous coronary interventions are performed. There has been, however, concerns of increased risk for clot formation in the heart arteries of patients treated with drug-eluting stents. Therefore, in order to lower the risk of clot formation, it is recommended that patients receiving these types of stents, be treated with dual antiplatelet therapy (blood thinning medication) for one year. The effect of this strategy, however, on clot formation and bleeding complications when utilizing "newer generation" stents, such as the Xience: Everolimus-eluting Stent, have not been well described.

Therefore, the aim of this registry study is to evaluate the risk of adverse cardiovascular events, including mortality, non-fatal myocardial infarction, stent thrombosis, hemorrhagic stroke, and severe bleeding in relation to the timing and discontinuation of dual antiplatelet therapy in patients treated with Xience drug-eluting stents, and compare it to patients that do not discontinue dual antiplatelet therapy.

DETAILED DESCRIPTION:
The introduction of drug-eluting stents (DES) into clinical practice is universally regarded as a revolutionary breakthrough in reducing the incidence of restenosis following percutaneous coronary intervention (PCI). The coating of stents with antiproliferative properties addresses a fundamental limitation of the earlier generation bare metal (uncoated) stents (BMS) - the in-growth of tissue through the struts of the stent that may eventually narrow the coronary artery resulting in recurrent ischemia. DES have greatly reduced the need for repeat revascularization, and thus, use of DES has rapidly become the de facto standard of care in the US.

The first two FDA-approved DES in the United States were the Cypher: Sirolimus-Eluting Coronary Stent and the TaxusExpress2™: Paclitaxel-Eluting Coronary Stent. Since then, the so-called 2nd generation DES which have come to market include the Xience: Everolimus-Eluting Coronary Stent and the Medtronic: Zotarolimus-Eluting Coronary Stent. Data from recent studies released in September of 2009 showed that Xience/Promus outperformed Boston's Taxus. Just prior to the release of this data, US market share was Xience 30%, Promus 24%, Taxus 22%, Endeavor 13%, and Cypher 11%. However, data was also released regarding Endeavor outperforming the Taxus stent as well, suggesting an upsurge is likely in US and world market share for Medtronic's Endeavor stent.

In the data recently presented from the SPIRIT IV trial, a randomized study between Xience and Taxus, significant benefits of Xience were found in comparison to the Taxus stent. There was a 38% reduction in target lesion failure and a 46% reduction in target lesion revascularization compared to Taxus. Notably, in this study of nearly 3700 patients, Xience had a low rate of stent thrombosis at 1-year of only 0.17%, compared to 0.85% for Taxus. The COMPARE study in higher-risk patients, also confirmed these results showing significant benefits of Xience V over Taxus Liberte at 1-year with regard to major adverse cardiac events and stent thrombosis.

These results suggest that there may be significant differences in outcomes favoring the use of 2nd generation DES, specifically as it relates to their superiority to 1st generation DES in reducing the need for repeat revascularization. There is, however, limited data examining the long-term safety of these devices when used in routine clinical practice. Furthermore, these DES have still not been fully studied in specific patient populations commonly encountered in routine clinical practice, including those with diabetes, chronic kidney disease, long-lesions, small vessels, and left main disease, among others. The outcomes revolve not only around efficacy of these stents in different clinical and angiographic scenarios, but also around the safety profiles. In particular, there has been great attention placed not only on the risk of stent thrombosis but also the timing of these events with the various DES, and how to reduce the incidence of them. The data available to date suggest favorable safety results for the Xience stent. However, in the ever changing world of dual antiplatelet therapy, and the duration of it, further understanding of these interactions are required. Currently, the majority of our efforts in reducing stent thrombosis have been channeled through more aggressive and longer duration of dual antiplatelet therapy. The effect of such strategies on other endpoints, such as bleeding complications after PCI, is unknown. These treatment strategies are based on our understanding of the need for dual antiplatelet therapy with 1st generation DES. Whether these same paradigms apply to 2nd generation DES, such as the Xience stent, is unclear. Furthermore, given that there continue to be significant questions regarding the precise rates of relatively rare clinical events, such as stent thrombosis and bleeding, strategies that allow us to estimate these rates when these devices are used in routine clinical practice, are warranted.

Specifically, the clinical impact of transient or permanent discontinuation of dual-antiplatelet therapy on these endpoints at various intervals after Xience implantation in routine clinical practice, has not been well characterized. As such, there continues to be considerable variability regarding the duration of dual antiplatelet therapy in routine clinical practice, regardless of the type of DES utilized. Therefore, a registry with rigorous long-term follow-up of patients treated with the Xience stent, that collects information on rare events, compliance with dual antiplatelet therapy, and relationships between use/non-use of dual antiplatelet therapy and adverse events would address these goals.

Accordingly, to better understand the long-term safety profile of the Xience stent in the overall population, as well as in those in whom dual antiplatelet therapy is discontinued, we propose to evaluate integrated patient data from the University of Pittsburgh Medical Center (UPMC) network system using two well-established institutions: the UPMC clinical sites and the University of Pittsburgh's Epidemiology Data Center (EDC). In brief, we propose to create the UPMC PCI-XIENCE registry, which will integrate the large-volume UPMC clinical sites with the well-established EDC as the data coordinating center. This will allow us to further investigate the long-term safety of the Xience stent as it is used in routine clinical practice.

Thus, the Specific Aims are to:

1. Evaluate the risk of stent thrombosis, hemorrhagic stroke, and severe bleeding in relation to the timing and discontinuation of dual anti-platelet therapy in patients treated with Xience drug-eluting stents.
2. Study the safety and efficacy of the Xience stent within specific understudied patient (diabetes mellitus, chronic kidney disease, women, minorities, etc) and angiographic (left main, bifurcation, saphenous vein graft, and small vessel disease) subgroups, among others.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing a coronary stenting procedure with the Xience drug-eluting stent
* Signed informed consent

Exclusion Criteria:

* Inability to sign informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of all consecutive patients who undergo coronary stenting with the Xience drug-eluting stent in any of the 4 University of Pittsburgh Medical Center's Hospitals (UPMC Presbyterian, UPMC Shadyside, UPMC Mercy, and UPMC Passavant).
Sampling Method: Non-Probability Sample
Enrollment: 2506 (Actual)
Dates: Start 2011-08; Primary Completion 2015-02 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Major Adverse Cardiovascular Events (MACE) | 24 months
  Combined end-point of all cause mortality, non-fatal myocardial infarction, stent thrombosis, need for repeat revascularization.

SECONDARY OUTCOMES:
Major Bleeding Events | 24 months
  A combined endpoint including subarachnoid hemorrhage, intracerebral hemorrhage, other/unspecified intracranial hemorrhage, gastric ulcer or gastrointestinal hemorrhage.

CONTACTS AND LOCATIONS:
Overall Officials: Oscar C Marroquin, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States